CLINICAL TRIAL: NCT04544371
Title: Evaluation of Gastric Residual Volume in Fasting Obese Patients Using Gastric Ultrasound: a Comparative Study
Brief Title: Ultrasound Assessment of Gastric Residual Volume in Obese Patients
Status: Completed | Type: Observational
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Atef Mohamed Sayed mahmoud, Principal investigator, Fayoum University Hospital
Other Study IDs: M420
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Aspiration Pneumonia
Keywords: Gastric residual volume; Obese; Ultrasound; Aspiration
MeSH Terms: conditions — Pneumonia, Aspiration; Obesity | interventions — Intubation, Gastrointestinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal weight patients: patients with body mass index =18-24.9 kg/m2 will be examined by abdominal ultrasound to assess gastric antrum cross sectional area in semi-sitting and right lateral positions
  Interventions: Device: gastric ultrasound; Procedure: nasogastric tube insertion
- obese patients: patients with body mass index >30 kg/m2 will be examined by abdominal ultrasound to assess gastric antrum cross sectional area semi-sitting and right lateral positions
  Interventions: Device: gastric ultrasound; Procedure: nasogastric tube insertion

INTERVENTIONS:
Device: gastric ultrasound — Focused gastric ultrasound was performed in semi-sitting position then right lateral position mindray curved transducer for examination of abdomen with low frequency (2-5 MHz) by a trained physician. The antrum of the stomach was located in the epigastrium after a sweep of the probe from left to right subcostal margins. This could be done using left lobe of liver as an anterior landmark and descending abdominal aorta as a posterior landmark
Procedure: nasogastric tube insertion — Nasogastric tube (18-french) was inserted after induction of anaesthesia and endotracheal intubation. Aspiration of gastric contents was performed through gentle suction using 50 ml syringe with synchronous epigastric massage and gentle movement of nasogastric tube in and out for 10 minutes after confirmation of nasogastric tube position.
  Other Names: Ryle tube

SUMMARY:
Gastric emptying is a major risk factor for aspiration of gastric contents.Aspiration into the lungs represents a fatal complication that can occur during anesthesia.

Not only gastric emptying importance to anesthetists is related to aspiration but also it is important to determine the systemic availability of substances given through the mouth. Delayed gastric emptying represents a major danger as it causes nausea and vomiting and prevents a return to oral feeding. Lastly it may cause morbidity and mortality.

Both humoral and neural influences have their impact on emptying. Volume and composition of gastric food act as major determinants for the rate of gastric emptying. The effect of body weight on gastric emptying are inconsistent.

ASA fasting guidelines application represents the primary method to avoid aspiration as it ensures that stomach is empty before induction of anesthesia.

These guidelines cannot be applied on all cases as in urgent or emergent situations or in morbidities associated with delayed gastric emptying.

Ultrasound can be used perioperatively to asses gastric content and volume at bedside.

DETAILED DESCRIPTION:
The objective of the current study is to evaluate gastric residual volume in obese patients versus healthy controls scheduled for elective surgery, using gastric ultrasound.

This prospective observational study was performed on 100 patients undergoing elective surgery from July 2019 to June 2020 at Fayoum University hospital after approval of the local institutional ethical committee (M420). A detailed informed consent was signed by the eligible participants before enrollment.

Our study adheres to the CONSORT guidelines. The study was conducted on 100 Patients were assigned to one of two groups of (50) patients in each group. Group obese ASA II from( 30-40) BMI, ASA III above 40 BMI without other comorbidities and group non obese ASA I control.Obese patients whose BMI >30 and healthy patients whose BMI = 18-24.9 who was scheduled for an elective surgery were included in this trial. All patients were enrolled in the study aged above >20 y. This study included patients scheduled for elective surgery after 8-hour overnight fast after a light meal.

Ultrasound scanning:

Focused gastric ultrasound by was performed by a trained physician in semi-sitting position then right lateral position using low frequency (2-5MHz) mindray curved transducer and mindray DP-20 ultrasound system. The antrum of the stomach was located in the epigastrium after a sweep of the probe from left to right subcostal margins. This could be done using left lobe of liver as an anterior landmark and descending abdominal aorta as a posterior landmark.

The antrum was considered to be empty if flat with juxtaposed anterior and posterior walls, fluid-containing if distended with thin walls and hypoechoic contents, solid -containing if distended with a content with mixed echogenicity according to antral shape and contents .

The antral cross sectional area (CSA) was measured using the two antral dimensions, craniocaudal (D1) and anteroposterior (D2) dimensions, according to the following equation: π [D1×D2]/4 provided that π = 22/7.

The gastric residual volume was calculated according to patient position as follows:

Bouvet and colleagues equation for semi-sitting position: gastric residual volume (ml) =215 + 57 log CSA (mm2) - 0.78 age (year) - 0.16 height (cm) - 0.25 weight (kg) - 0.80 ASA.

Perlas and colleagues equation for right lateral position: gastric residual volume (ml) = 27.0 + 14.6 × right-lateral CSA - 1.28 × age.

Using the classification of Ven de Putte and perlas, the study could asses the risk of aspiration as follows: (a) low risk of aspiration: patients with empty antrum and patients with gastric residual volume less than 1.5 ml/kg.(b) high risk of aspiration: patients with solid contents and patients with gastric residual volume more than 1.5 ml/kg.

Nasogastric tube (18-french) was inserted after induction of anaesthesia and endotracheal intubation. Aspiration of gastric contents was performed through gentle suction using 50 ml syringe with synchronous epigastric massage and gentle movement of nasogastric tube in and out for 10 minutes after confirmation of nasogastric tube position.

Statistical Analysis The collected data were organized, tabulated and statistically analyzed using SPSS software statistical computer package version 22 (SPSS Inc, USA). Numerical variables were not normally distributed and were presented as median and interquartile range (IQR); Mann-Whitney U test was used as a test of significant. Qualitative data were presented as numbers and percentages, and the chi-squared test was used to determine significance. A two-sided P-value of <0.05 was considered statistically significant.

Sample size Sample size calculated using G-Power© software version 3.1.7 results with effect size (0.57), two sided (two tails) type I error 0.05 and power of 80%, each group should include at least (50) Subjects. the authors expected no dropout rates or missing data.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged from 20 years to 60 years
* Patients scheduled for elective surgery after an 8-hour overnight fast after a light meal (200 ml milk, 50 g white cheese, and 120 g bread).
* American society of anesthesiologists physical status I-III.

Exclusion Criteria:

* Pregnancy
* Renal failure
* Liver cell failure
* History of upper GIT morbidity (hiatus hernia and gastric cancer)
* History of upper abdominal surgery.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This prospective observational study will be performed on 100 patients undergoing elective surgery in fayoum university
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
measurement of gastric residual volume in semi-sitting position | 5 minutes preoperatively
  in cubic centimetre

SECONDARY OUTCOMES:
measurement of gastric residual volume in right lateral position. | 5 minutes preoperatively
  in cubic centimetre
Antral cross sectional area in semi-sitting position | 5 minutes preoperatively
  in millimetre square
Antral cross sectional area in right lateral position | 5 minutes preoperatively
  in millimetre square
volume of fluid aspirated from nasogastric tube | 1 minute after induction of anesthesia
  in cubic centimetre
grade of aspiration risk | 5 minutes preoperatively
  less (low risk) or more (high risk) 1.5 millilitre/kilogram
Grading for assessment of antrum of the stomach | 5 minutes preoperatively
  : 3 points as follows: grade 0: empty antrum, grade 1: minimal fluid in right lateral position only, grade 2: distention of antrum in both right lateral and semi-sitting position

OTHER OUTCOMES:
Age | 1 hour preoperatively
  in years
Weight | 1 hour preoperatively
  in kilograms
Body mass index | 1 hour preoperatively
  in kilograms/ square metre
Height | 1 hour preoperatively
  in centimetre

CONTACTS AND LOCATIONS:
Overall Officials: Atef M sayed, MD, Principal Investigator — Fayoum University; maged L Bolis, MD, Study Chair — Fayoum University
Locations (1):
- Fayoum University hospital, El Fayoum Qesm, Faiyum Governorate Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sun H, Wu CW, Zhang D, Makay O, Zhao Y, Carcofaro P, Kim HY, Dionigi G, Pino A, Caruso E, Pontin A, Pappalardo V. New Paradigms for Neural Monitoring in Thyroid Surgery. Surg Technol Int. 2019 May 15;34:79-86. PMID 30664223
- [Background] Bakalinis E, Makris I, Demesticha T, Tsakotos G, Skandalakis P, Filippou D. Non-Recurrent Laryngeal Nerve and Concurrent Vascular Variants: A Review. Acta Med Acad. 2018 Nov;47(2):186-192. doi: 10.5644/ama2006-124.230. PMID 30585070
- [Background] Neelakanta G, Chikyarappa A. A review of patients with pulmonary aspiration of gastric contents during anesthesia reported to the Departmental Quality Assurance Committee. J Clin Anesth. 2006 Mar;18(2):102-7. doi: 10.1016/j.jclinane.2005.07.002. PMID 16563326
- [Background] Bouvet L, Mazoit JX, Chassard D, Allaouchiche B, Boselli E, Benhamou D. Clinical assessment of the ultrasonographic measurement of antral area for estimating preoperative gastric content and volume. Anesthesiology. 2011 May;114(5):1086-92. doi: 10.1097/ALN.0b013e31820dee48. PMID 21364462
- [Background] Zaremba S, Shin CH, Hutter MM, Malviya SA, Grabitz SD, MacDonald T, Diaz-Gil D, Ramachandran SK, Hess D, Malhotra A, Eikermann M. Continuous Positive Airway Pressure Mitigates Opioid-induced Worsening of Sleep-disordered Breathing Early after Bariatric Surgery. Anesthesiology. 2016 Jul;125(1):92-104. doi: 10.1097/ALN.0000000000001160. PMID 27171827